CLINICAL TRIAL: NCT06186193
Title: Mind Your Pain: Validating the Mindful Interoceptive Exposure Task (MIET) for Patients With Chronic Low Back Pain
Brief Title: Mind Your Pain: Validating a Mindful Interoceptive Exposure Task for Patients With Chronic Low Back Pain
Acronym: MyP
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 20-32001; U19AR076737 (NIH)
Record Dates: First submitted 2023-12-06; First posted 2023-12-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Chronic Low-back Pain
Keywords: chronic low back pain; interoceptive exposure; attention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mindful Interoceptive Exposure: Mindful Interoceptive Exposure Phone-based interoceptive exposure task as attention exercise with chronic low back pain
  Interventions: Behavioral: MyP

INTERVENTIONS:
Behavioral: MyP — see above: attention exercise based on phone app
  Other Names: Mind your Pain

SUMMARY:
The usual coping mechanism with chronic pain is distraction, It is unclear whether the opposite, sensory monitoring, can benefit patients with chronic low back pain (cLBP). The study assesses the feasibility and acceptability of a 2-minute phone-based attention exercise, used several times a day over 8 weeks plus a 1-hour introduction, in patients with cLBP. The attention exercise is based on mindfulness-based interoceptive exposure, a task that has been tested before in a mixed pain population in Australia.

DETAILED DESCRIPTION:
Mind your Pain (MyP), also known as Mindfulness-based Interoceptive Exposure Therapy (MIET) is an innovative brief mindfulness-based task, developed within the frame of mindfulness-based cognitive therapy, and has been pilot tested in a small cohort of 15 patients with chronic musculoskeletal pain, the majority with cLBP, in Australia. It consists of an individual guided 1-hour introduction session and a 1 to 2-minute attention task subsequently performed several times per day over 12 weeks. The task will be provided by a smart phone app and be sent to participants as phone message reminders at up to 5 times per day: according to participant preference once in the morning and once at bedtime, as well as up to 3 additional times when participants are asked to use the app whenever they perceive the pain at its worst. The task is to focus on the most intense pain sensation in a detached and equanimous way and carefully observe potential changes in five aspects of that sensation: space (region/ borders/ immobile/ moving); sense of mass (heavy/ neutral/ light), temperature (cold/ warm/ hot/ neutral); density (dense/ solid/ loose/ constricted), and borders (diffuse/ sharp). This neutral sensory-descriptive interoceptive attention focus is aiming at preventing the learned aversive response to pain that entails ruminating thoughts, and negative affect rather than immediate sensory awareness. The pilot study in 15 chronic pain patients showed significant beneficial pre-post effects (Cohen's d, ES) of 0.96 for pain anxiety, 0.86 for pain duration and 1.37 for pain intensity, maintained at 2-month follow-up. The investigators offer the MyP-MIET to patients in the US with clearly defined chronic low back pain over 8 weeks, validate it with 30 participants for feasibility and acceptability and exploratory self-report key pain outcomes and objectively (using QST and fMRI), who fit a low interoceptive awareness phenotype. The investigators also use qualitative exit interviews.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic low back pain (cLBP) defined according to the NIH Research Task Force recommendation on Research Standards for cLBP: pain at least half the days in the past 6 months, by using 2 questions and a human figure drawing illustrating the region as the space between the lower posterior margin of the rib cage and the horizontal gluteal fold.
2. Average pain in the last month at least 3 out of 10 on Numeric Rating Scale [range 0 - 10, for 0 signifying no pain and 10 signifying worst pain imaginable]. This level of pain allows comparability of the study results with the majority of cLBP studies. Pain rated less than 3 is too mild to detect improvement.
3. Men and women aged 18-65 years old. We are not enrolling younger children as they are not part of the Intensive Pain Rehabilitation Therapy program. 65 is our upper limit for age due to changes in blood flow on the MRI.
4. Eligibility will be assessed using the following questions: "(1) How long has back pain been an ongoing problem for you? and (2) How often has low-back pain been an ongoing problem for you over the past 6 months?" A response of greater than three months to question 1, and a response of "at least half the days in the past 6 months" to question 2 would meet the cLBP eligibility criterion.
5. Ability to speak English. We do not have the capacity, given the resources available in this proposal, to translate all course material and conduct groups into another language. We have previously enrolled Hispanic participants into other studies who were fluent in English, and expect to do this in the proposed study.
6. Low level of interoceptive awareness and habitual distraction as coping mechanism with pain. This is defined as:

   1. MAIA summary score below the population mean score of 3.41. The value of 3.41 is the mean value of a sample of primary care patients at Kaiser Permanente in a prior study.
   2. the MAIA Non-Distraction score is below 2.91 [possible range 0-5]. The value of 2.91 is the mean value plus standard deviation in the same sample.4 This eligibility criterion was chosen to test the hypothesis that the MIET task will be able to increase interoceptive awareness in patients with chronic low back pain with below average interoceptive awareness and preference for distracting themselves from their pain experience.
7. Owning a smart phone: the task is smart phone-based.

Exclusion Criteria:

1. Unable to provide informed consent.
2. A substance abuse, mental health, or medical condition that, in the opinion of investigators, will make it difficult for the potential participant to participate or that may need immediate changes in medical management that will affect study outcome measures. Such conditions may include cancer, liver failure, renal failure, pain conditions from inflammatory diseases (e.g. rheumatoid arthritis, ankylosing spondylitis, lupus), malignancies or abdominal aortic aneurysm, muscle weakness from radiculopathy. Radiculopathy or sciatic pain is NOT excluded as long as the condition is stable and does not lead to significant movement restrictions or <4/5 muscle weakness. Persons with significant substance abuse or mental health conditions that interfere with social functioning may be disruptive. Oher medical or mental health conditions that need immediate changes in management need to be addressed before starting the study so that more reliable baseline measurements can be made. Patients who may need assessment for potentially necessary surgical interventions may not be able to complete the study. Regular opioid prescription is not an exclusion if stabile over the past 3 months.
3. Spine related current or history of spine infection, spine tumor, vertebral fracture, cauda equina syndrome. Colorblindness or left handedness. Conditions would increase heterogeneity of the sample.
4. Blindness, severe vision problems, deafness, severe hearing problems, bipolar or manic depression and not taking medication, major depression, psychoses (major), a substance abuse condition, dementia, unable to get up and down from the floor. Condition might make it difficult to participate.
5. Some other serious medical conditions that may alter key study outcomes, including untreated hypothyroidism, renal failure, and cirrhosis. Conditions that may alter key study outcomes.
6. Involvement in a lawsuit related to their back. Complicated medico-legal issues that could lead to individuals having a financial incentive to not report improvement.
7. Involved in Worker's Compensation claim.
8. Pregnant, breast-feeding, or planning to get pregnant in the next 12 months or less than 3 months post-partum. Particular back problems than may be associated with pregnancy and delivery may confound study outcomes.
9. Lack of stable housing or plan to move out of the area within the next 6 months.
10. MRI-related exclusion criteria: Cardiac pacemaker, metal fragments in eyes/skin/body (shrapnel), subjects who have ever been a metal worker/welder; history of eye surgery/eyes washed out because of metal, aortic aneurysm clips, prosthesis, by-pass surgery/coronary artery clips, hearing aid, heart valve replacement, subjects with an I.U.D, a shunt (ventricular or spinal), electrodes, metal plates/ pins/screws/wires, or neuro/bio-stimulators (TENS unit), vision problems uncorrectable with lenses, claustrophobia; inability to lie still on one's back for approximately 60 minutes; prior neurosurgery; older tattoos with metal dyes; unwillingness to remove nose, ear or face jewelry, braces or permanent dental retainers. Iron-containing metal parts in the body can potentially be dislocated by strong magnetic fields and preclude assessment with MRI.
11. Received a steroid or botox injection in or near the spine in the last 3 months. This may alter key study outcomes.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with chronic low back pain living in the Bay Area
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2023-07-21 (Actual)

PRIMARY OUTCOMES:
app usage | daily over 8 weeks
  acceptability/feasibility: number of app uses
Pain, Enjoyment of life and General activity scale (PEG) | pre-post 8 weeks
  scale range is 0-30, higher scores are worse outcome. change in PEG scores for combined pain intensity and pain interference
Numeric Rating Scale (NRS) for pain intensity in the past 7 days. Range 0-10, with 10 worst pain. | past 7 days
  pain intensity

SECONDARY OUTCOMES:
Quantitative Sensory Testing (QST), pain threshold to thermal stimulus | pre-post 8 weeks
  QST measures pain threshold with a heat stimulus in a pain physiology laboratory.
resting state functional Magnetic Resonance Imaging (rsfMRI) | pre-post 8 weeks
  rsfMRI assesses the structural integrity of the brain and detects changes in grey cortical thickness in distinct brain areas. Reduced thickness indicates less neural density.
fMRI connectivity | pre-post 8 weeks
  Using a thermal stimulus in the MRI scanner, changes from before to after the intervention in fMRI connectivity between distinct brain areas can be detected.
Multidisciplinary Assessment of Interoceptive Awareness (MAIA) | pre-post 8 weeks
  This is an 8-scale instrument, each ranging 0-5, with higher scores indicating higher interoceptive awareness, in order to assess pre-post changes.

CONTACTS AND LOCATIONS:
Overall Officials: Wolf E Mehling, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco; Osher Center for Integrative Health, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data Depository all IPD on which the main publication is based on
Supporting Information: Study Protocol
Time Frame: May 2024
Access Criteria: To be determined

REFERENCES:
- [Derived] Mehling WE, Strigo IA, Goldman V, Hartogensis W, Adler SR, Lotz J, Hecht FM. Mind your pain: A single-arm feasibility study to assess a smartphone-based interoceptive attention training for patients with chronic low back pain. PLoS One. 2024 Oct 24;19(10):e0307690. doi: 10.1371/journal.pone.0307690. eCollection 2024. PMID 39446767